CLINICAL TRIAL: NCT05980806
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Selinexor Monotherapy in Subjects With JAK Inhibitor-naïve Myelofibrosis and Moderate Thrombocytopenia
Brief Title: A Study of Selinexor Monotherapy in Subjects With JAK Inhibitor-naïve Myelofibrosis and Moderate Thrombocytopenia
Acronym: SENTRY-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-MF-044
Record Dates: First submitted 2023-07-24; First posted 2023-08-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Myelofibrosis; Moderate Thrombocytopenia; Mild Thrombocytopenia
Keywords: Myelofibrosis; Selinexor; Total Symptom Score; Myelofibrosis Symptom Assessment Form; Spleen Volume Reduction; TSS50; SVR35; JAK2; KPT-330; Pacritinib; Ruxolitinib; Momelotinib; Thrombocytopenia; Abs-TSS
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocytopenia | interventions — selinexor; ruxolitinib; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selinexor 60 mg (Arm 1) (Experimental): Participants will receive selinexor 60 milligrams (mg) oral tablets once weekly (QW) (Days 1, 8, 15, and 22 of each 28-day cycle) until PD, intolerable toxicity, or until they meet the criteria for discontinuation of study treatment. Optional add-on medication dosing may be initiated based on Spleen Volume Reduction (SVR) values at Week 12 or Week 24 of treatment.
  Interventions: Drug: Selinexor 60 mg; Drug: Ruxolitinib; Drug: Pacritinib; Drug: Momelotinib
- Selinexor 40 mg (Arm 2) (Experimental): Participants will receive selinexor 40 mg oral tablets QW (Days 1, 8, 15, and 22 of each 28-day cycle) until PD, intolerable toxicity, or until they meet the criteria for discontinuation of study treatment. Optional add-on medication dosing may be initiated based on Spleen Volume Reduction (SVR) values at Week 12 or Week 24 of treatment.
  Interventions: Drug: Selinexor 40 mg; Drug: Ruxolitinib; Drug: Pacritinib; Drug: Momelotinib

INTERVENTIONS:
Drug: Selinexor 60 mg — Participants will receive selinexor 60 mg oral tablets QW.
  Other Names: KPT-330
  Arms: Selinexor 60 mg (Arm 1)
Drug: Selinexor 40 mg — Participants will receive selinexor 40 mg oral tablets QW.
  Other Names: KPT-330
  Arms: Selinexor 40 mg (Arm 2)
Drug: Ruxolitinib — Participants will receive ruxolitinib per local package insert.
  Other Names: JAKAFI
Drug: Pacritinib — Participants will receive pacritinib per local package insert. For countries where not approved, 200 mg twice daily is the starting dose.
  Other Names: VONJO
Drug: Momelotinib — Participants will receive momelotinib per local package insert.
  Other Names: OJJAARA

SUMMARY:
The main purpose of this study is to evaluate the efficacy of selinexor in JAKi-naïve participants with myelofibrosis (MF) and with normal platelet counts or with mild to moderate thrombocytopenia based on spleen volume reduction (SVR). Additional efficacy and safety parameters will also be assessed during the study.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of MF or post-ET or post-PV MF according to the 2016 World Health Organization (WHO) classification of MPN, confirmed by the most recent local pathology report
* Measurable splenomegaly during the screening period as demonstrated by spleen volume of greater than or equal to (>=) 450 cubic square centimeter (cm^3) by MRI or CT scan (results from MRI or CT imaging performed within 28 days prior to C1D1 are acceptable)
* DIPSS risk category of intermediate-1 with symptoms, or intermediate-2, or high-risk
* ECOG Performance Status less than or equal to (<=) 2
* Platelet count of greater than or equal to (>=) 50 x 10^9/L without platelet transfusion within 7 days prior to the first dose of selinexor
* Absolute neutrophil count (ANC) >=1.0 × 10^9/L without need for growth factors within 7 days prior to the first dose of selinexor
* Adequate liver function as defined by the following: aspartate transaminase (AST) and alanine transaminase (ALT) <= 2.5 × upper limit normal (ULN) and serum total bilirubin <= 3×ULN
* Calculated creatinine clearance (CrCl) greater than (>) 15 milliliter per minute (mL/min) based on the Cockcroft and Gault formula
* Active symptoms of MF as determined by presence of at least 2 symptoms with an average score >= 5 or total score of >= 12 at screening (at least 5 of 7 consecutive days immediately preceding C1D1) using the MFSAF V4.0
* Must provide bone marrow biopsy samples (samples obtained up to 3 months prior to C1D1 are permitted) at screening and during the study
* Currently not eligible for stem cell transplantation
* Must be willing to complete the MFSAF V4.0 daily during the study for evaluating the symptom response (i.e., TSS50)

Key Exclusion Criteria:

* More than 10% blasts in peripheral blood or bone marrow (accelerated or blast phase)
* Previous treatment with JAK inhibitors for MF
* Previous treatment with selinexor or other XPO1 inhibitors
* Females who are pregnant or lactating
* Prior splenectomy, splenic radiation, or a splenic embolization within 6 months prior to C1D1
* History of myocardial infarction, unstable angina, percutaneous transluminal coronary angioplasty (PTCA), coronary artery bypass graft (CABG), cerebrovascular accident (transient ischemic attack [TIA]), ventricular arrhythmias, congestive heart failure class > 2 per New York Heart Association (NYHA) within 6 months of C1D1
* Unable to tolerate two forms of antiemetics prior to each dose for the first two cycles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Spleen Volume Reduction ≥35% (SVR35) at Week 24 | At Week 24
  Measured by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) Scan by Investigator assessment.

SECONDARY OUTCOMES:
Absolute Mean Change in Total Symptom Score (Abs-TSS) from baseline to Week 24 | At Baseline and Week 24
  Measured by the Myelofibrosis Symptom Assessment Form (MFSAF) V4.0.
Incidence and severity of TEAEs, including TRAEs and SAEs | From Baseline to EoS (approximately 48 months)
  Measured by the NCI CTCAE Grading Scale, v. 5, as assessed and graded by the Investigator

CONTACTS AND LOCATIONS:
Locations (70):
- United States (7):
  - City of Hope - Duarte Main Site, Duarte, California
  - Maryland Oncology Hematology - Independent of SCRI/ US Oncology, Columbia, Maryland
  - Weill Cornell Medicine NewYork-Presbyterian, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment Sveti George - Base 1, Plovdiv
  - University Hospital Sv.Ivan Rilski - Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases - EAD Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD Department of Clinical Hematology, Stara Zagora
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada
- Fakultní nemocnice Olomouc, Olomouc, Czechia
- Aarhus Universitetshospital, Aarhus N, Central Jutland, Denmark
- France (8):
  - Institut Bergonié, Bordeaux, Aquitaine
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Tours, Hôpital Bretonneau Service d'Hématologie thérapie cellulaire, Tours, Indre-et-Loire
  - Chu De Nîmes - Institut De Cancérologie Du Gard, Nîmes, Occitanie
  - Centre Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Hôpital Saint-Louis, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Priest-en-Jarez
- Germany (2):
  - Marien Hospital Düsseldorf, Düsseldorf
  - University Hospital Jena, Jena
- Greece (5):
  - Laiko General Hospital of Athens, Athens, Attica
  - University General Hospital Attikon, Athens, Attica
  - "Georgios Papanikolaou" General Hospital of Thessaloniki, Thessaloniki, Central Macedonia
  - University General Hospital of Ioannina, Hematology Department, Ioannina, Epirus
  - University General Hospital of Larissa, Hematology Department, Larissa, Thessaly
- Semmelweis Egyetem, Budapest, Hungary
- Israel (3):
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
- Italy (11):
  - Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, Milan
  - Hematology Division, Mauriziano Hospital, University of Turin, Orbassano, Torino
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino, Turin
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori - IRST, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Università Campus Bio-Medico di Roma, Rome
- Spaarne Gasthuis, Hoofddorp, Netherlands
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - AIDPORT, Skórzewo
  - Medicover Clinical Integrated Systems Sp. z o.o., Torun
- Romania (3):
  - Coltea - Spital Clinic, Bucharest
  - Spitalul Filantropia - Craiova, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
- South Korea (4):
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seocho, Seoul
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital, Busan
- Spain (8):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital San Pedro de Alcantara, Cáceres
  - Institut Català d'Oncologia Girona, Girona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan District
- Guy's and Saint Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided